CLINICAL TRIAL: NCT00177996
Title: Pharmacotherapy in Depression With Panic Spectrum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Andrea Fagiolini, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 010403
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Major Depression
Keywords: depression; anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertaline high dose titration (Active Comparator): The study was a double-blind study in which subjects diagnosed with major depression complicated by lifetime panic spectrum symptomatology were randomized to either high (but still within the standards of normal clinical practice) or low dose titration schedules of Sertraline hydrochloride. The doses and titration schedules used in this arm (Sertaline high dose titration) are consistent with recommended FDA guidelines.
  Interventions: Drug: sertraline hydrochloride
- Sertaline low dose titration (Active Comparator): The study was a double-blind study in which subjects diagnosed with major depression complicated by lifetime panic spectrum symptomatology were randomized to either high (but still within the standards of normal clinical practice) or low dose titration schedules of Sertraline hydrochloride. The doses and titration schedules used in this arm (Sertaline low dose titration) are consistent with recommended FDA guidelines.
  Interventions: Drug: sertraline hydrochloride

INTERVENTIONS:
Drug: sertraline hydrochloride — The study was a double-blind study in which subjects diagnosed with major depression complicated by lifetime panic spectrum symptomatology were randomized to either high (but still within the standards of normal clinical practice) or low dose titration schedules of sertraline. The doses and titration schedules used in this study are consistent with recommended FDA guidelines.
  Other Names: sertraline hydrochloride low versus high dose titration

SUMMARY:
This research study is being conducted to find out if certain individuals benefit from taking medication for their depression with a low dose of the antidepressant medication Zoloft.

DETAILED DESCRIPTION:
Researchers at the University of Pittsburgh Medical Center Health System are currently recruiting men and women, ages 18 to 60, to examine the effectiveness of the FDA-approved medication sertraline (Zoloft) for major depression.

Participants will be randomly assigned to one of two groups. Each group will begin and continue taking Zoloft at different doses. A physician will follow eligible participants weekly for approximately 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18-60;
* Current diagnosis of major depression, and a rating of ³15 on the HRS-D-25; - -Presence of significant, co-existing panic-agoraphobic spectrum symptoms,
* Absence of ongoing therapy with psychotropic medications (except for intermittent use of nonbenzodiazepine hypnotics) or willingness to be withdrawn from an ineffective ongoing antidepressant medications
* Physically healthy,
* Female participants of childbearing potential must be practicing a medically acceptable form of double-barrier birth control or using oral contraceptives such as birth control pills, implants, or injections;

Exclusion Criteria:

* Females who are pregnant or breast-feeding;
* History of suicide attempt in the 6 months prior to entry, active suicidal ideation, or significant suicide risk;
* History of hypersensitivity to or current use of sertraline;
* Unstable or untreated medical conditions,
* Participants who do not wish to discontinue current, ineffective antidepressant treatment;
* Participants who have recently begun psychotherapy (less than 3 months prior to study entry);
* Diagnosis of current panic disorder, psychosis, substance or alcohol abuse, anorexia, bulimia, dissociative, bipolar disorder, or any other psychiatric or medical illness that would interfere with the best treatment strategy for the potential participant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2001-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Somatic Symptoms Scale (SSC) | 1 week
  Scale to evaluate somatic and panic like symptoms

SECONDARY OUTCOMES:
Hamilton Rating Scale For Depression- 25 item (HRSD 25) | 1 week
  scale to evaluate depressive symptoms
Global Assessment of Functioning (GAF) | past week
  scale to evaluate ability to function

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Fagiolini, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Insititue and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided